CLINICAL TRIAL: NCT04491058
Title: Assessment of Subsynovial Connective Tissue Thickness in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Elise Robben, Principal investigator, KU Leuven
Other Study IDs: S63134
Record Dates: First submitted 2020-07-14; First posted 2020-07-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Subsynovial Connective Tissue; Ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Carpal tunnel syndrome patients: Subjects with unilateral or bilateral carpal tunnel syndrome
  Interventions: Diagnostic Test: SSCT thickness measurement
- Healthy: Subjects without carpal tunnel syndrome
  Interventions: Diagnostic Test: SSCT thickness measurement

INTERVENTIONS:
Diagnostic Test: SSCT thickness measurement — Thickness measurement with ultrasound

SUMMARY:
The general aim of this research is to gain insight in the role of SSCT in the etiology and progression of CTS. We hypothesize that (degenerative) damage of the SSCT occurs early on in the pathogenesis of CTS. Fibrotic damage to the SSCT will lead to altered morphology and biomechanical characteristics. This eventually may lead to damage of the median nerve. To examine the SSCT an ultrasound technique described by Van Doesburg et al. 2012 will be used First, the reliability of the US technique to characterize morphology of the SSCT will be investigated. Secondly, cross-sectional data will be collected in healthy subjects and CTS patients to provide descriptive parameters and to describe differences between patients and controls. In the final part a prospective study will be conducted to look at changes of SSCT thickness over time and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* For CTS patients
* Human adults, 18 years and older
* Complaints compatible with CTS (Katz Hand Diagram[31] rating of 'classic', 'probable' or 'possible' or typical clinical signs)
* Indication for electrodiagnostic testing
* Informed consent to participate
* For Healthy subjects
* Human adults, 18 years and older
* Negative electrodiagnostic testing and scoring 'unlikely' at Katz Hand diagram
* Informed consent to participate

Exclusion Criteria:

* Pregnancy
* History of renal disease, diabetes, chemotherapy, tumors, other neurological diseases (e.g., polyneuropathy), thyroid disease
* Problems of the upper limb, e.g., degenerative and inflammatory joint disease, gout, tendinopathy at the wrist, acute trauma of the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with and without carpal tunnel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Inter- and intrarater reliability of subsynovial connective tissue thickness measurement with ultrasound | baseline
  To determine whether ultrasound is a reliable tool to measure SSCT thickness in patients with carpal tunnel syndrome and healthy subjects.
Baseline subsynovial connective tissue thickness | Baseline
  To determine correlations between SSCT thickness and participant characteristics (e.g., age, gender) in patients with carpal tunnel syndrome and healthy subjects. To obtain normative data for SSCT thickness in healthy subjects and patients with carpal tunnel syndrome.
Change in subsynovial connective tissue thickness after 3, 6 and 12 months | 3, 6, 12 months
  To evaluate the change in SSCT thickness over time in patients with carpal tunnel syndrome and healthy subjects (without intervention).
Change in subsynovial connective tissue thickness after treatment | 3, 6, 12 months
  To evaluate the effect of treatment (i.e., surgery or infiltration) on SSCT thickness in patients with carpal tunnel syndrome. Orthopedic surgeon decides independently if and which treatment is necessary for the patient. If possible, to subgroup patients according to the correlation between their response to treatment, assessed with electrodiagnostic testing and clinical variables, and (change in) SSCT thickness.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No